CLINICAL TRIAL: NCT04659551
Title: Engaging the Immune System to Improve the Efficacy of Neoadjuvant Chemo-endocrine Therapy for Premenopausal Luminal B Breast Cancer Patients
Brief Title: Neoadjuvant Chemo-endocrine Therapy and Immunotherapy for Pre-menopausal Luminal B Breast Cancer Patients
Acronym: GIADA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIADA Trial; 2016-004665-10 (EudraCT Number)
Record Dates: First submitted 2018-02-23; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Triptorelin Pamoate; exemestane; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Epirubicin 90 mg/mq + Cyclophosphamide 600 mg/mq i.v. every 3 weeks for 3 courses, followed by Nivolumab (240 mg flat dose i.v. each 2 weeks) for 8 courses plus exemestane 25 mg (orally, continuous daily dose, to be continued until surgery). LHRH analogue (Triptorelin 3.75mg 1 fl i.m. every 28 days) started concomitantly to anthracycline based chemotherapy, to be continued until surgery.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Triptorelin; Drug: Exemestane; Drug: Nivolumab

INTERVENTIONS:
Drug: Epirubicin — Epirubicin 90 mg/mq i.v. every 3 weeks for three cycles
Drug: Cyclophosphamide — Cyclophosphamid 600 mg/mq i.v. every 3 weeks for three cycles
Drug: Triptorelin — Triptorelin 3.75 mg i.m. every 4 weeks until surgery
Drug: Exemestane — Exemestane 25 mg oral continuous daily dose until surgery
Drug: Nivolumab — Nivolumab 240 mg flat dose i.v. every two weeks for 8 cycles
  Other Names: BMS-936558

SUMMARY:
Multicentric, phase II neoadjuvant trial in hormone-positive, HER-negative, luminal B, premenopausal breast cancer patients stage II-IIIA. Patients receive as neoadjuvant treatment before surgery: three courses of anthracycline-based chemotherapy followed by exemestane p.o. daily plus nivolumab i.v. 2-weekly for 8 courses. GnRH analogues are started concomitantly with chemotherapy and maintained until the completion of neoadjuvant treatment.

DETAILED DESCRIPTION:
This is a multicenter, phase II neoadjuvant trial in hormone-sensitive, HER-negative, luminal B, premenopausal breast cancer patients stage II-IIIA.

Patients will undergo a core-biopsy of the primary tumor, for the histological diagnosis and the biological characterization of the tumor.

After confirmation of eligibility and informed consent signature, the patients will start neoadjuvant treatment including:

Epirubicin 90 mg/mq + Cyclophosphamide 600 mg/mq i.v. every 3 weeks for 3 courses, followed by the combination of Nivolumab (240 mg flat dose i.v. each 2 weeks) for 8 courses and exemestane 25 mg (orally, continuous daily dose, to be continued until surgery). Patients will start LHRH analogue (Triptorelin 3.75mg 1 fl i.m. every 28 days) concomitantly to anthracycline-based chemotherapy, to be continued until surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they met all the following criteria

* age >18 yrs
* female patients
* ECOG Performance Status 0-1
* must have signed and dated an IRB/IEC-approved written informed consent form in accordance with regulatory and institutional guidelines before the performance of any protocol-related procedures
* Primary diagnosis of invasive breast cancer, HR positive (ER ≥ 10% and/or PgR ≥10% by IHC) and HER2 negative (IHC 0/1+ and/or FISH/CISH negative) according to local assessment.
* Histologic grade 3 and/or Ki67 >20% according to local assessment.
* Stage II-IIIA
* Eligible for neoadjuvant chemotherapy according to multidisciplinary evaluation.
* Premenopausal status
* Normal organ and marrow function
* Availability of tumor tissue suitable for biological and molecular examination before starting primary treatment
* Ability to understand and willingness to sign a written informed consent document

Exclusion criteria:

Patients will be excluded from the study for any of the following reasons

* Stage IIIB, IIIC, and inflammatory breast cancer
* Stage IV breast cancer
* Prior treatment with chemotherapy, biologic therapy, endocrine therapy or radiotherapy for the treatment of the newly-diagnosed breast cancer.
* Contraindication to anthracycline-based chemotherapy.
* Received any investigational treatment within 4 weeks of study start.
* Any other concurrent chemotherapy, biologic therapy, endocrine therapy or radiotherapy for cancer treatment.
* Known HIV, HBV, HCV infection or any positive tests for HBV and HCV indicating acute or chronic infection.
* Known severe hypersensitivity to any of the study drugs or excipients or known severe hypersensitivity reactions to monoclonal antibodies.
* Major surgical procedure or significant traumatic injury within 28 days prior to treatment initiation or anticipation of need for major surgery during the course of study treatment.
* History of allogenic organ transplantation
* Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident /stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of treatment initiation.
* Subjects with active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Any other serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a subject's ability to comply with the study requirements, substantially increase risk to the subject, or impact the interpretability of study results.
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
* Lack of physical integrity of the upper gastrointestinal tract, clinically significant malabsorption syndrome, or inability to take oral medication.
* Psychiatric illness/social situations that would limit compliance with study requirements
* Subjects assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol
* Current pregnancy and/or lactation.
* Refusal to adopt adequate (highly effective) contraception methods.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
pathological complete response (pCR) | up to 7 months from enrolment
  ypT0ypN0

SECONDARY OUTCOMES:
clinical objective response | up to 6 months from enrolment
  cOR
molecular response | up to 7 months from enrolment
  Ki67
Breast conserving surgery | up to 7 months from enrolment
  Surgery type
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 100 days from last nivolumab dose
  Adverse Events
Correlative biomarkers | Tumor samples will be collected at baseline, at 14 days after completion of anthracycline-based chemotherapy (about 7 weeks after first dose of Epirubicin), at surgery (about 30 weeks after first dose of Epirubicin)
  correlation between different biomarkers expression at baseline and pathological response

CONTACTS AND LOCATIONS:
Overall Officials: Pierfranco Conte, MD, Principal Investigator — University of Padova
Locations (5):
- Italy (5):
  - Arcispedale S. Anna, Cona, FE
  - Centro di Riferimento Oncologico di Aviano (CRO), Aviano, PN
  - Azienda Ospedaliera Universitaria di Parma, Parma, PR
  - Arcispedale S. Maria Nuova, Reggio Emilia, RE
  - Istituto Oncologico veneto IRCCS, Padua

REFERENCES:
- [Derived] Dieci MV, Guarneri V, Tosi A, Bisagni G, Musolino A, Spazzapan S, Moretti G, Vernaci GM, Griguolo G, Giarratano T, Urso L, Schiavi F, Pinato C, Magni G, Lo Mele M, De Salvo GL, Rosato A, Conte P. Neoadjuvant Chemotherapy and Immunotherapy in Luminal B-like Breast Cancer: Results of the Phase II GIADA Trial. Clin Cancer Res. 2022 Jan 15;28(2):308-317. doi: 10.1158/1078-0432.CCR-21-2260. Epub 2021 Oct 19. PMID 34667023